CLINICAL TRIAL: NCT06636435
Title: A Phase I, First in Human Study of CBA-1205, Anti-DLK1 Monoclonal Antibody in Patients With Advanced Solid Tumors.
Brief Title: A Phase I, First in Human Study of CBA-1205, Anti-DLK1 Monoclonal Antibody in Patients With Advanced Solid Tumors, Hepatocellular Carcinoma (HCC), Melanoma, and Pediatric Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chiome Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 1205-001; jRCT2080225288 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-09-30; First posted 2024-10-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors; Hepatocellular Carcinoma (HCC); Malignant Melanoma; Pediatric Cancer
Keywords: DLK1; First in human; Phase I; Antibody; solid tumor; Hepatocellular Carcinoma; CBA-1205; Melanoma; Pediatric Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Melanoma; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- CBA-1205: Part 1 (Experimental): CBA-1205 injection is administered at 2-week intervals in seven cohorts (0.1, 0.3, 1, 3, 10, 20, 30 mg/kg) in patients with solid tumor.
  Note: In the study treatment period, CBA-1205 is intravenously administered at 2-week intervals in a 28-day cycle.
  Interventions: Drug: CBA-1205 Part 1
- CBA-1205: Part 2 (Experimental): CBA-1205 (20, 30 mg/kg) injection is administered at 2-week intervals in 28-day cycles in patients with HCC .
  Note: The study drug is administered at 2-week intervals until any of the criteria for discontinuation of study treatment are met.
  Interventions: Drug: CBA-1205 Part 2
- CBA-1205: Part 3 (Experimental): CBA-1205 injection is administered at 2-week intervals in 28-day cycles in patients with HCC.
  Note: The study drug is administered at 2-week intervals until any of the criteria for discontinuation of study treatment are met.
  Interventions: Drug: CBA-1205 Part 3
- CBA-1205 : Part 4 (Experimental): CBA-1205 injection is administered at 2-week intervals in 28-day cycles in patients with Malignant Melanoma.
  Note: The study drug is administered at 2-week intervals until any of the criteria for discontinuation of study treatment are met.
  Interventions: Drug: CBA-1205 Part 4
- CBA-1205: Part 5 (Experimental): CBA-1205 injection is administered at 2-week intervals in 28-day cycles in patients with Pediatric Cancer.
  Note: The study drug is administered at 2-week intervals until any of the criteria for discontinuation of study treatment are met.
  Interventions: Drug: CBA-1205 Part 5

INTERVENTIONS:
Drug: CBA-1205 Part 1 — CBA-1205: 0.1, 0.3, 1, 3, 10, 20, 30 mg/kg (Intravenous solution)
  Arms: CBA-1205: Part 1
Drug: CBA-1205 Part 2 — CBA-1205: 20 mg/kg and 30 mg/kg (Intravenous solution)
  Arms: CBA-1205: Part 2
Drug: CBA-1205 Part 3 — CBA-1205: 30 mg/kg (Intravenous solution)
  Arms: CBA-1205: Part 3
Drug: CBA-1205 Part 4 — CBA-1205: 20 mg/kg (Intravenous solution)
  Arms: CBA-1205 : Part 4
Drug: CBA-1205 Part 5 — CBA-1205: 10 mg/kg (The initial cohort, Intravenous solution)
  Arms: CBA-1205: Part 5

SUMMARY:
In this first-in-human, muticenter, non-randomized, open-label, standard 3+3 dose escalation Phase I study encompasses 5 parts (Part 1-5). The purpose of this FIH study is to evaluate the safety and tolerability profile of CBA-1205.

DETAILED DESCRIPTION:
To evaluate safety and efficacy of CBA-1205 in the following five parts in a stepwise manner:

Part 1

* In Part 1, safety and tolerability in patients with Solid Tumor where no standard treatment is available, or who are intolerable or non-responder to the standard treatment will be evaluated. Initial dose for Part 2 will be determined.

Part 2

* In Part 2, safety and tolerability in patients with advanced and/or recurrent Hepatocellular Carcinoma which are unresectable, or who are intolerable or non-responder to the standard treatment will be evaluated. Recommended dose in this population will be determined.

Part 3

* In Part 3, safety and efficacy at the recommended dose in patients with advanced and/or recurrent Hepatocellular Carcinoma which are unresectable, or who are intolerable or non-responder to the standard treatment will be evaluated.

Part 4

* In Part 4, safety and efficacy in patients with Malignant Melanoma who are refractory or intolerant to standard therapy.

Part 5

* In Part 5, safety, tolerability and the recommended dose of the study drug in patients with Pediatric Cancer where no standard treatment is available, or who are intolerable or non-responder to the standard treatment will be evaluated.

PK analysis

ELIGIBILITY:
Inclusion Criteria:(Part 1-4)

* Patients who provide voluntary written informed consent to participate in the study
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of≤1
* Patients with preserved renal function as evidenced by laboratory data obtained within 7 days before enrollment (creatinine: ≤ ULN ×1.5)
* Patients who meet the following laboratory criteria of bone marrow function as evidenced by laboratory data obtained within 7 days before enrollment: Neutrophil count;≥1500/μL, Platelet count; ≥75000/μL, Hemoglobin;≥9.0 g/dL.
* Patients having Solid Tumors with no standard therapy available or refractory or intolerable to standard therapy (Part2, 3)
* Patients with Child-Pugh A or B (Part2, 3)
* Patients with Malignant Melanoma who are refractory or intolerant to standard therapy (Part 4)

Inclusion Criteria:(Part 5)

* Patients who provide voluntary written informed consent to participate in the study from both the subject (if aged 16 years or older) and their legal representatives
* Japanese patients aged 2 years or older and under 20 years at the time of informed consent
* Patients with a Lansky Performance Status (LPS) of ≥70 (for patients aged 15 years or younger) or a Karnofsky Performance Status (KPS) of ≥70 (for patients aged 16 years or older)
* Patients with preserved renal function as evidenced by laboratory data obtained within 7 days before enrollment (eGFR ≥60 mL/min/1.73 m²)
* Pediatric patients with cancers with no standard therapy available or refractory or intolerable to the standard therapy

Exclusion criteria: (Part1-5)

* Patients who have undergone major surgery within 28 days before enrollment
* Patients who have received anticancer treatment with surgical therapy, radiation therapy, and/or drug therapy within 14 days before enrollment
* Patients who have received anticancer treatment with immune checkpoint inhibitor, etc. within 28 days before enrollment
* Patients with Grade 2 or higher concurrent disease or prior therapy-related toxicity
* Patients who have received any other investigational product within 28 days before enrollment
* Patients with current or previous inadequately controlled or clinically significant cardiac disease
* Patients who, in the opinion of the investigator or subinvestigator, is not appropriate

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Part 1, 2 and 5 - Dose limiting toxicity : For 28 days after the first dose of study treatment
  DLTs are assessed according to CTCAE v.5.0 during the first cycle (28 days).
Adverse Event | Adverse event : Maximum 12 months
  An adverse event is any untoward or unintended sign, symptom, or disease in a subject administered an investigational product, whether or not it is related to the investigational product

SECONDARY OUTCOMES:
Serum CBA-1205 concentration | From Day 1 to Day 43 (or until Discontiuation of treatment)
  Blood samples are collected to assess the serum concentration of CBA-1205.
Immunogenicity | From Day1 to Day 43 (or until Discontiuation of treatment)
  Blood samples are collected to assess the serum anti-CBA-1205 antibody.
Efficacy | Screening, Day 1 of Cycle 2 and 3, and Day 1 of even-numbered cycles from Cycle 4 onward until treatment discontinuation. Maximum 12 months
  Antitumor response evaluated in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
  Tumor markers

OTHER OUTCOMES:
Exploration of biomarkers: | Baseline through disease progression assessed (Maximum 12 months.)
  Exploration of biomarkers:
  Delta-like 1 homolog (DLK1)-related marker

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - National Cancer Center Hospital, Chūō, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakamura K, Takahashi K, Sakaguchi I, Satoh T, Zhang L, Yanai H, Tsukumo Y. A Novel Glycoengineered Humanized Antibody Targeting DLK1 Exhibits Potent Anti-Tumor Activity in DLK1-Expressing Liver Cancer Cell Xenograft Models. Int J Mol Sci. 2024 Dec 19;25(24):13627. doi: 10.3390/ijms252413627. PMID 39769389
- [Background] Katsuya Y, Ikeda M, Koyama T, Sato J, Okada M, Matsubara N, Kondoh C, Mukohara T, Watanabe K, Kotani D, Ogawa Y, Taoka S, Yamamoto N. A Phase I, First-In-Human Study of CBA-1205, an Anti-DLK1 Monoclonal Antibody, in Patients With Advanced Solid Tumors. Cancer Sci. 2025 Apr;116(4):1012-1022. doi: 10.1111/cas.16454. Epub 2025 Jan 20. PMID 39832211
- See also: Sponsor Page — https://www.chiome.co.jp/?id=en